CLINICAL TRIAL: NCT06931353
Title: Effect of the Anticholinergic Drug Burden on Postoperative Delirium in Elderly Chinese Patients: A Nested Case-Control Study
Acronym: ADB and POD
Status: Completed | Type: Observational
Sponsor: Hao Li (Other)
Responsible Party: Sponsor-Investigator, Hao Li, associate chief physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: ChinaPLAGH-ADB and POD
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Delirium - Postoperative
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to investigate the association between preoperative anticholinergic drugs burden and postoperative delirium in elderly Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* patients over 65 years; Undergoing general anesthesia; Inpatients who had surgery between Aprill 1, 2020 and Aprill 1, 2022.

Exclusion Criteria:

* ASA grade V; preoperative Mini-Mental State Examination (MMSE) score <24;history of neurological disorders (such as cerebrovascular disease or dementia); emergency surgeries; operative duration ≤30 minutes, and cases with >5% missing data.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients over 65 years
Sampling Method: Non-Probability Sample
Enrollment: 10536 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
postoperative delirium | 7 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- First Medical Center of Chinese PLA General Hospital, Beijing, China